CLINICAL TRIAL: NCT00688948
Title: A Pilot Study Looking At The Use Of Alfuzosin In The Treatment Of Bladder Dysfunction In Patients With Multiple Sclerosis
Brief Title: Alfuzosin for Voiding Dysfunction in Multiple Sclerosis (MS)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Jerzy B Gajewski MD, Capital District Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RS/2007-035; JBGMS01
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-02

CONDITIONS: Multiple Sclerosis; Bladder Dysfunction
Keywords: pilot clinical trial
MeSH Terms: conditions — Multiple Sclerosis | interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin — Alfuzosin 10 mg once daily po for 12 weeks
  Other Names: Xatral

SUMMARY:
Multiple Sclerosis is often associated with severe functional deficits resulting in a range of progressive impairments. Approximately 80% of patients have bladder symptoms at the time of diagnosis and up to 97% will have bladder symptoms during the course of the disease. To date, the vast majority of treatment has been centered on the use of medications to control "bladder spasms" and the use of catheters to help patients empty the bladder. There have been very few studies looking at medications like Alfuzosin that may help in controlling bladder symptoms in Multiple Sclerosis. Alfuzosin has been shown to significantly improve voiding symptoms and bladder emptying in patients with prostatic enlargement. There have been no controlled studies yet to determine whether this treatment helps patients with Multiple Sclerosis. The purpose of this study is to determine if Alfuzosin improves bladder symptoms and quality of life in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
OBJECTIVE The primary objective of this study is to evaluate the use of Alfuzosin in the treatment of bladder dysfunction in patients with Multiple Sclerosis (MS).

STUDY POPULATION Twenty (20) participants aged 18 years of age who have been diagnosed with Multiple Sclerosis and lower urinary tract symptoms will be treated with Alfuzosin.

DESIGN This is a single institution, non-randomized, non-blinded pilot study of the use of Alfuzosin in the treatment of bladder dysfunction in MS patients. After the initial screening visit patients will be given 10 mg of Alfuzosin to be taken daily once daily.

STUDY INSTRUMENTS The primary end points of this study are a reduction in the ICIQ questionnaires and improvement in uroflow, post-void residual (PVR) and voiding diaries. All patients will have a detailed history and physical examination at the beginning of the study and at 12 weeks follow-up. Women will have a pregnancy test at the beginning of the study. Participants will be given the ICIQ questionnaires, uroflow and PVR at the screening visit and at week 6 and 12. In addition, these patients will be asked to maintain a three day voiding diary prior to week 2 and week 12. Assessments for safety (blood pressure and heart rate) will be collected at baseline and at the last visit. Blood tests will be performed to check for liver, kidney and prostate problems at the baseline visit. Adverse events will be recorded at all visits and when spontaneously reported by the study participants.

DURATION OF STUDY The study will be 12 weeks in duration.

ELIGIBILITY:
Inclusion Criteria:

1. Participant should be eighteen years of age or older.
2. Participant should have LUTS secondary to Multiple Sclerosis as defined below.
3. Participant should have frequency ≥ 8/day and/or incontinence and/or nocturia ≥ 2/night and/or urgency and/or urinary retention.
4. Participant should be able to understand, speak and read English.
5. Participant 's urine culture should not show any evidence of urinary tract infection.
6. Participant should be willing to take part in the study and sign the consent form.
7. Female participants consents to use a medically acceptable method of birth control throughout the entire study period and for four weeks after the study is completed. Medically acceptable methods of contraception that may be used by the study participants and/or their partner includes abstinence, birth control pills or patches, diaphragm with spermicide, IUD, condom and vaginal spermicide, surgical sterilization, vasectomy, progestin implants or injections.

Exclusion Criteria:

1. Participant with known hypersensitivity to Alfuzosin.
2. Participant with history of postural hypotension and/or syncope.
3. Participant has used another alpha blocker within the last 30 days.
4. Participant has active urethral stricture disease.
5. Participant has a history of prostate cancer within the preceding five years.
6. Participant has hepatic dysfunction.
7. Participant has renal dysfunction.
8. Participant has unstable angina pectoris.
9. Participant has a positive pregnancy test at the time of screening.
10. Participant has a history of serious social, mental or medical conditions that would stop patient from taking part in the study.
11. Participant has a history of alcohol or drug abuse within the last five years.
12. Participant who is currently being treated for chronic bacterial prostatitis or painful bladder syndrome/interstitial cystitis.
13. Participant has a significant medical problem which the investigator considers a serious risk for the patient to be part of the study.
14. Use of any investigational drug or device within the last 6 months.
15. Participant who is unwilling or unable to abide by the requirements of study.
16. Participant has a bladder infection proven by urine culture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy measures will be the ICIQ-LUTSqol questionnaire, the IPSS questionnaire, uroflow/PVR and the voiding diaries. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy B Gajewski, MD, Principal Investigator — QEII Health Science Centre
Locations (1):
- QE II Health Science Centre, Halifax Infirmary, Halifax, Nova Scotia, Canada